CLINICAL TRIAL: NCT05390372
Title: Efficacy of Breast Milk in Healing of Skin Damage Due to Tape Peeling in Premature Babies: A Randomized Study
Brief Title: Efficacy of Breast Milk in Healing of Skin Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayse Sonay Turkmen, Prof.Dr, Prof.Dr, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Humanmilk
Record Dates: First submitted 2022-05-11; First posted 2022-05-25 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Milk Expression, Breast
MeSH Terms: conditions — Breast Milk Expression | interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- humanmilk (Experimental): For skin damage care of preterm newborns randomly assigned to the breast milk group, their own breast milk will be applied topically once every 60 minutes until complete healing. Skin damage in newborns will be evaluated by an independent nurse and specialist doctor for 60 minutes during the treatment, and the score will be given and recorded. A minimum decrease of 1 point in the skin condition assessment scale score will be considered to indicate 'improvement'. The decision that the skin integrity of the newborn is completely healed will be made by the neonatal doctor independent of the trial. Areas between 0-3 on the newborn skin condition assessment scale will be considered healed. Breastfeeding does not have any side effects in preterm newborns.
  Interventions: Other: human milk
- routine care group (Experimental): cream applied as part of hospital routine practice
  Interventions: Other: Routine care group

INTERVENTIONS:
Other: human milk — For skin damage care of preterm newborns randomly assigned to the breast milk group, their own breast milk will be applied topically once every 60 minutes until complete healing. Skin damage in newborns will be evaluated by an independent nurse and specialist doctor for 60 minutes during the treatment, and the score will be given and recorded. A minimum decrease of 1 point in the skin condition assessment scale score will be considered to indicate 'improvement'. The decision that the skin integrity of the newborn is completely healed will be made by the neonatal doctor independent of the trial. Areas between 0-3 on the newborn skin condition assessment scale will be considered healed. Breastfeeding does not have any side effects in preterm newborns.
  Arms: humanmilk
Other: Routine care group — cream applied as part of hospital routine practice
  Arms: routine care group

SUMMARY:
The population of the research will be preterm infants born 35-36 weeks of gestation, hospitalized in the Neonatal Intensive Care Unit of Karaman State Hospital, whose skin is damaged due to Intravenous (IV) vascular access fixation bands, and whose skin has not been subjected to any other application before. Calculation of the sample number of the research; It was determined that at least 24 newborns should be assigned to each group (α = 0.05 and β = 0.19) to show that the 1 degree difference between the cream group and the breast milk group was significant for 80.7% strength. It is planned to take a premature baby. As data collection tools, Premature Babies Descriptive Information Form, Newborn Skin Condition Assessment Scale, Medical Adhesives and Solvents Used in the Neonatal Intensive Care Unit, Human Milk and routine care will be used.

DETAILED DESCRIPTION:
Randomization The process of inclusion of newborns into groups will be randomly assigned using the computer program (https://www.randomizer.org). Which letter will be the breast milk or routine care group was determined by the closed opaque envelope method at the beginning of the study. Accordingly, the letter A will be used for the breast milk group and the letter B will be used for the cream group. According to the black bag drawn randomly by an independent nurse from the research, which group it will be in will be determined.

Hypotheses H1: The use of topical breast milk is more effective than the routine care in the healing of skin damage due to tape stripping, which is used in the detection of IV vascular access in premature babies.

H2: The use of routine care is more effective than topical breast milk in the healing of skin damage due to tape stripping, which is used in the detection of IV vascular access in premature babies.

Variables of the Study Dependent variables: Scores from the newborns' "Neonatal Skin Condition Assessment Scale".

Independent variables: Sociodemographic characteristics, two different methods including breast milk and routine care.

Data Collection Tools Information Form for Premature Babies It consisted of questions including information about the gender, gestational week, current weight, birth weight, postnatal age, length of hospitalization, and nutritional status of the premature newborns included in the study.

Newborn Skin Condition Rating Scale It is a measurement tool developed by Lund and Osborne (2004) to evaluate the skin condition of term, premature or post-term, healthy or sick newborn babies. Turkish validity and reliability of the scale Calisir et al. (2016) with 96 newborn babies who were hospitalized in Adnan Menderes University Neonatal Intensive Care Unit and selected using the improbable method. The scale consists of three items and each item includes an evaluation criterion. These are respectively dryness, erythema and deterioration of skin integrity/peeling. Each item of the scale, which was developed as a three-point Likert scale, gets points from 1 to 3. The lowest score that can be obtained from the scale is 3 and the highest score is 9, and a high total score indicates that the newborn's skin condition is bad.

Medical Adhesives and Solvents Used in the Neonatal Intensive Care Unit Adhesives in the form of fabric, silk, polyester, paper, plastic, foam, polyurethane film used in neonatal intensive care. It is used to fix IV routes. It is recommended not to use adhesive tape solvents because of the dangers of toxicity in absorption and skin irritation in premature skin. Silk plaster is used in the neonatal intensive care unit, which is included in the research, and isotonic liquid is used as tape solvent.

Routine care: The routine care, which is routinely used in the treatment of tape stripping in the neonatal intensive care unit, will be used within the scope of the research. Features of the routine care used routinely by the clinic: It can be used in children from birth. The cream has no known contraindications. The cream is applied to the lesioned area of the skin as a thin layer. Instructions for proper use and dose/frequency of administration: Cream; It is applied to the lesioned area several times a day. There is no time limit on the use of the cream.

Research Implementation Plan Preliminary Application of the Research; In the research; In order to evaluate the effects of breast milk and routine care on the healing of skin damage due to tape peeling, pre-treatment will be applied to 4 preterm newborns in the newborn intensive care unit of Karaman Training and Research Hospital. Thus, the difficulties in the application of the methods were determined in advance and it was planned to eliminate these problems by the researcher.

First Stage;

* Newborns to be included in this study receive care and treatment in an incubator because they are hospitalized in the neonatal intensive care unit.
* The follow-up and follow-up of the newborn's skin evaluation at all stages of this study will be followed and evaluated by the physician of the neonatal intensive care unit.
* The silk patch used in the IV catheter fixation of the newborn will be slowly removed by the neonatal nurse parallel to the skin. In order to facilitate the removal of the plaster, the plaster will be removed slowly and carefully with cotton moistened with isotonic liquid, softening the tape.
* In the first stage, a nurse and a specialist doctor who are independent of the study will evaluate the skin damage caused by the removal of intravenous vascular access in preterm newborns by using the "Neonatal Skin Condition Assessment Scale" by the observers, and the score will be given and recorded.
* Alcohol-free cotton wipes dipped in water will be used to clean the damaged skin area of newborns in both groups.
* Preterm newborns will be randomly assigned to 2 groups as breast milk and routine care group.

Second Stage;

Breast Milk Group:

For skin damage care of preterm newborns who are randomly assigned to the breast milk group, their own breast milk will be applied topically once in 60 minutes until complete healing. A decrease of at least 1 point in the condition assessment scale score will be considered to indicate 'improvement'. The decision that the skin integrity of the newborn is completely healed will be made by the neonatal doctor independent of the trial. Areas between 0-3 on the newborn skin condition assessment scale will be considered healed. Breastfeeding does not have any side effects in preterm newborns (Qu-Yang et al., 2013; Rosali et al., 2015; Rodrigues et al., 2017).

Routine Care Group:

For skin damage care of preterm newborns who are randomly assigned to the cream group, the cream will be applied topically once in 60 minutes until complete healing. A reduction of 1 point will be considered to indicate 'improvement'. The decision that the skin integrity of the newborn is completely healed will be made by the neonatal doctor independent of the trial. Areas between 0-3 on the newborn skin condition assessment scale will be considered healed.

In both groups, skin damage will be evaluated once before the procedure and 10 times after the procedure (with an interval of one hour), a total of 11 times.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal consent of the parents,
* The newborn is less than 37 weeks of gestation,
* Being in the Neonatal Intensive Care Unit,
* The intravenous catheter has been fixed to the skin with a silk patch,
* For intravenous catheter fixation, the bands remain on the skin for a minimum of 24 hours and a maximum of 32 hours,
* While removing the adhesive tape, remove it slowly and carefully by softening the tape with cotton moistened with water,
* The parent speaks and understands Turkish comfortably,
* Stable health status
* Having spontaneous breathing
* Not being exposed to a painful procedure at least half an hour before the interventions.
* Not taking opioid or non-opioid analgesics
* Not receiving any antibiotic treatment,
* Having breast milk

Exclusion Criteria:

* Parent's inability to speak and understand Turkish easily,
* Parents do not give written and verbal consent,
* Intravenous catheter not fixed to the skin with a silk patch,
* For intravenous catheter fixation, the bands should not remain on the skin for a minimum of 24 hours and a maximum of 32 hours,
* Removal of the intravenous catheter from the skin using a solvent solution,
* Having ventilator support
* Presence of congenital anomaly
* Using analgesic / narcotic analgesic drugs
* Receiving any antibiotic treatment,
* Continuous sedative treatment
* Discontinuation of topical breast milk or cream application procedure for any reason
* Parent's wish to leave the study

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — preterm newborns
Enrollment: 36 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
skin damage | 3 weeks
  The change in skin damage after the intervention with newborn skin condition assessment scalewill be monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayşe Sonay Türkmen, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No